CLINICAL TRIAL: NCT07360821
Title: Investigation of Autonomic Stress Response Patterns in College Students With Varying Physical Activity Levels
Acronym: ANS Stress/PA
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025601H; 2025601H (Other: Beijing sport university)
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autonomic Nervous System Activity; Cardiovascular; Physical Activity Level
Keywords: SKNA; HRV; Blood Pressure Variability; Athletes; Cardiopulmonary Exercise Testing
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sedentary Control: Healthy adults with minimal physical activity, screened via SBQ and IPAQ-S questionnaires as baseline controls
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing
- Endurance Athletes: Long-distance runners or triathletes with over 1 year of regular aerobic training (e.g., 800m+ running, swimming).
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing
- Strength Athletes: Athletes specializing in anaerobic/power-based training, such as weightlifting, wrestling, or sprinting.
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing
- Traditional Ethnic Sports: Practitioners of mind-body exercises like Tai Chi or Baduanjin, emphasizing respiratory control and mild intensity
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing — Cardiopulmonary Exercise Testing (CPET) is a non-invasive, integrated assessment of the cardiovascular, respiratory, and muscular systems' responses to physical stress.

SUMMARY:
This study aims to investigate the differences in cardiovascular stress response patterns among individuals with various physical activity levels (sedentary controls and different types of athletes). By synchronously monitoring ECG, heart rate, skin sympathetic nerve activity (SKNA), blood pressure, and cardiac output, the study will characterize physiological dynamics during resting, orthostatic challenge, cold pressor stress, and maximal exercise.

DETAILED DESCRIPTION:
Participants will be categorized into five groups based on their training background: sedentary, endurance, strength, technical, and traditional ethnic sports. The experimental protocol includes baseline measurements in lying, standing, and sitting positions, followed by a series of acute stress tests: a lie-to-stand orthostatic test, a slow breathing test, and a cold pressor test. Finally, participants will perform a ramp incremental exercise test on a cycle ergometer. Synchronous physiological data including HRV and SKNA will be collected to evaluate the dynamic regulation of the autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

Healthy young adults aged 18-25 years

Body Mass Index (BMI) within the range of 18.5-23.9 kg/m 2

No history of systematic professional athletic training (for sedentary group) or confirmed training background (for athlete groups)

No exercise contraindications or history of cardiovascular, respiratory, or metabolic diseases

No family history of sudden cardiac death

Ability to understand the study protocol and sign the informed consent form

Exclusion Criteria:

History of limb sports injury within the past 6 months or unhealed fractures

Habits of smoking or chronic alcohol consumption

Presence of implanted electronic devices (e.g., pacemakers)

Clinical diagnosis of psychiatric disorders such as anxiety or depression

Recent use of medications affecting autonomic or cardiovascular function

Regular practice of meditation or ongoing psychotherapy

Irregular menstrual cycles (for female participants)

Peripheral neuropathy or other autonomic nervous system disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of 60-80 healthy adult volunteers (college students). Participants are categorized into five distinct groups based on their habitual physical activity levels and training backgrounds: 1) Sedentary controls, 2) Endurance athletes, 3) Strength athletes, 4) Technical athletes, and 5) Traditional ethnic sports practitioners (e.g., Tai Chi). Gender balance is maintained across all groups.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Baseline (10-minute rest), during the 10-minute mental stress test, and during the cardiopulmonary exercise test (approx. 20 minutes)
  Time-domain metrics (e.g., RMSSD, SDNN) derived from ECG recordings to evaluate cardiovagal modulation and cardiac autonomic balance.
Skin Sympathetic Nerve Activity | Baseline (10-minute rest), during the 10-minute mental stress test, and during the cardiopulmonary exercise test (approx. 20 minutes)
  Integrated average SKNA (aSKNA) and burst metrics measured via surface electrodes to assess sympathetic nerve firing

IPD SHARING:
Plan to Share IPD: Undecided